# Informed Consent for participation in a Clinical Study

# "Detection of Coronary Artery Calcifications by whole blood Transcriptome analyzed by Artificial InTelligence algorithms. (CAC-TRAIT study)"

Esteemed patient,

We invite you to participate in a clinical study to be conducted at Clínica Sagrada Familia, owned by ROSARIO DEL PLATA S.A., CUIT 30-67769850-7, located at José Hernández 1642, CABA (the "Center"), under the sponsorship and organization of MULTIPLAI TANGO SAS (the "Sponsor"), and under the leadership of Study Principal Investigator Dr. Santiago Miriuka <a href="mailto:santiago@multiplaihealth.com">santiago@multiplaihealth.com</a> and Center Principal Investigator Dr Gastón A. Rodriguez Granillo +54 011 4014 6000.

It is the Sponsor's concern to seek better ways to diagnose and treat heart disease and your contribution to this end will be appreciated. You are invited to participate in this study either because you have to undergo a chest CT scan for a medical indication, or because your physician wishes to estimate your coronary artery calcium score.

Your participation is strictly voluntary, and you may refuse to participate in the study without prejudice, as well as withdraw from the study at any time you wish. Furthermore, your participation does not entail any change to the treatments that have been previously agreed upon with your primary care physician.

Clinical studies are fundamental for the advancement of medicine and the understanding of diseases. In order to achieve these goals, it is necessary to conduct clinical trials with the voluntary participation of patients. To do so, patients must be informed of the scope and risks of their participation, and sign an informed consent form that supports their decision to be part of it. Please read the following paragraphs carefully to understand the study, and then you will have the opportunity to discuss it with one of the investigators to answer any questions you may have. Finally, if you agree, please sign this consent form meaning that:

- You understand the scope of the study and the procedures to be performed.
- You are ready and willing to participate in the study.
- You know and your rights to participate in this study have been explained to you.
- You understood the form and purposes for which your personal data will be processed.

#### 1 What does the clinical study consist of?

The objective of the Study Sponsor is to develop a diagnostic method for the detection of cardiovascular disease by means of a blood test. To do this, a blood sample is taken to

analyze its RNA (a subtype of DNA) and another sample is taken to perform a clinical analysis (blood glucose, cholesterol, hematocrit, etc.). A buccal swab is then performed in order to obtain a DNA sample.

The results of the analysis will be used by the Sponsor to train an artificial intelligence algorithm to differentiate which of the samples carry the genetic information of the disease and which do not.

At the end of the follow-up study, it will also be explored whether the genetic information contained in the blood sample differs between participants who eventually developed a cardiovascular event (e.g., heart attack, stroke) and those who did not.

#### What are the procedures to be performed during the development of the study?

The blood collection procedure for RNA analysis is very simple, as you must donate only 2.5 milliliters of blood (¼ of the usual amount drawn during a routine clinical analysis). The collection is performed from a peripheral vein using a standard technique. The RNA from your blood will be sent to a Sponsor laboratory located in the United Kingdom for analysis, as no such studies are performed in the United Kingdom. The second blood draw (clinical analysis) will be 10 ml and is performed following the same procedure. This sample will be sent to Stamboulian Laboratory, a local clinical analysis laboratory owned by CENTRO DE ESTUDIOS INFECTOLÓGICOS SACEI, or to another local clinical analysis laboratory to be designated in the future that meets industry standards. The third procedure consists of a cheek and gum swab for the collection of a cell sample to obtain DNA. In all cases, care will be taken to ensure that the samples submitted do not contain data that would allow third parties to identify you and/or link that RNA sample to you. The fourth procedure consists of a non contrast gated cardiac CT by ECG ("coronary calcium score").

Once the blood and saliva have been donated and the chest CT scan has been performed, an interviewer from the Center will call you by telephone once a year and ask you a series of questions about your health status. If, during the time of the study (5 years), you have any health-related problems, an investigator authorized by the Center for such purposes will collect that information from your medical records or other available source document (epicrisis).

#### 3 What are the risks of my participation in the study?

The risks to your health are minimal, as the blood draw is the one that is routinely performed. Complications of this procedure are rare, and may consist of transient pain at the drawing site or the formation of a local hematoma. Rarely, more serious complications such as thrombophlebitis or local infection may occur. To reduce this complication, the blood sample will be drawn by a technician trained in this procedure.

Cheek swabbing involves obtaining the sample by rubbing a buccal swab against the inside of the cheeks and gums, and poses no risk to your health.

ECG-triggered non-contrast cardiac CT ("coronary calcium score") is based on X-ray imaging. The X-rays present in the CT scan pass through the body to produce images of internal structures such as the heart or lungs. All living beings are continuously exposed

to radiation from natural sources. For example, in the United States, the average person receives an effective radiation dose of about 3 mSv per year from the environment (from naturally occurring radioactive materials and solar radiation). In this study, you will receive a total effective radiation dose of between 1 and 1.5 mSv (compared to a dose of approximately 7 mSv in a conventional chest CT scan), so the risk of radiation-associated complications is virtually nonexistent (0.05 in 1000).

By signing this Informed Consent you do not waive your rights under the Civil and Commercial Code, and Argentine laws regarding civil liability for damages. In case of damage, injury or adverse event related to the study and you are covered by PRUDENCIA Compañía Argentina de Seguros Generales S. A. under policy number 00178983 - Contact: 0800-345-0085. If you have any questions about your participation in this study or in case of any discomfort related to the study, you may contact Dr. Gastón A. Granillo at telephone +54 011 4014 6000.

#### 4. Does my participation in the study bring me any benefits?

Every participant in the study will receive a written return (Report) from the Center's investigators with information provided by the Sponsor on the presence and extent of coronary artery calcifications, which is useful as a tool for cardiovascular prevention. You will be able to provide this report to your primary care physician. The information obtained from this study will allow in the future to improve the early detection of future diseases. You will not receive any reports or returns regarding the DNA-RNA determinations made in the framework of the study.

#### 5. What categories of my Personal Data will be processed and for what purposes?

5.1 For the purpose of your participation in the study, the following categories of data will be collected:

### 5.1.1 Identifying data:

- Full name
- ID
- Sex
- Address
- Contact data (e-mail and telephone)
- 5.1.2. Medical Data: Data collected or inferred from the procedures detailed in point 2 of this document, and from any interview conducted within the framework of the study by the Center's physicians.
  - 5.1.3. Pseudonomization of the Data: For the purposes of conducting the study, it is intended that your Identifying Information and Medical Data will be handled pseudonymously, using a coding mechanism so that third parties other than the Center and/or the Center's investigators cannot identify you or associate you and your Identifying Information with the Medical Data obtained in connection with the study. Whenever the Center or the Sponsor sends your Medical Data to any other entity involved in the conduct of any activity related to this study, it will do so in a

pseudonymized form. In this sense, the treatment of your Identifying Information that we call "pseudonymization" implies that access to it will be protected at all times by passwords, only accessible to the Center and/or the Center's Investigators, but not to the Sponsor or any other entity or third party.

In this sense, your Identifying Data will only be included at the time of recruitment in a form kept separately from the rest of the study by the Center, and coded, and only for the purpose of follow-up by the Center.

- 5.2. The purposes for which your Personal Data will be collected and processed are:
- 5.2.1. Processing of Identifying Data: This data will be collected and processed by the Center for the following purposes:
- - Storage, treatment and conservation for the registration of the participants of the study by the Center, and to be able to receive and evacuate consultations from the participants as well as requests for access, updating, rectification or suppression of personal data by the participants and holders of personal data.
- To provide participants with the Report containing information provided by the Sponsor on the presence and extent of coronary artery calcifications, which is useful as a tool for cardiovascular prevention.
- Follow-up of the participants and be able to contact them to interview them and ask questions about the participant's health status, within the framework of the study and always with the purposes of the study as indicated herein.
- Collect and process the information from the interviews with the participants, and enter it into the participant's clinical history and other available source documents (epicrisis).
- Collect and process interview information and share the results of the interviews with the Sponsor or such entities as the Sponsor may direct the Center to share, in a pseudonymized manner and for the purposes stated herein.
- To comply with the obligations of storage, treatment and conservation of the data of the participants of medical studies, for the terms and by virtue of the legal obligations of the Center in relation to the applicable regulations.
- 5.2.2. Processing of Pseudonymized Medical Data: This data will be collected and processed by the Center, the Sponsor and/or other entities involved in the study for the following purposes:
- Storage, processing and preservation for the Sponsor's health-related medical-scientific research and analysis purposes.
- -- Storage, treatment and conservation for legal purposes of the Center and to be able to receive and evacuate consultations of the participants as well as requests of access, update, rectification or suppression of personal data on the part of the participants and holders of personal data.

- Sponsor's medical-scientific research to develop better ways to detect, diagnose and treat cardiovascular diseases, by means of blood and other sample analysis.
- Sponsor's medical-scientific research to train artificial intelligence algorithms or other technologies developed or to be developed in the future, with the objective of differentiating which of the samples carry the genetic information of cardiovascular disease and which do not, and also to train artificial intelligence algorithms or other technologies developed or to be developed in the future, for other purposes of detection, diagnosis and treatment of diseases in general.
- Collaboration of the Sponsor with the Center's Researchers with the Reports to be delivered to the participants on the presence and extent of coronary artery calcifications, which is useful as a tool for cardiovascular prevention.
- Collaborate with the Center's Investigators in the elaboration of follow-up interviews of the participants and any other reports to be delivered to the participants.
- Validate results obtained through experts and/or technologies developed or to be developed in the future.
- Elaborate and present scientific-medical reports and/or publications on the topics addressed by the study, or its results, as well as on other related topics.
- Elaborate new medical-scientific research questions or processes.
- Sponsor's medical-scientific research to train artificial intelligence algorithms or other technologies developed or to be developed in the future, related to health that may or may not be used and/or patented and/or commercialized by Sponsor or third parties.

#### 6. How is your Pseudonymized Health Information shared?

In order to fulfill the purposes detailed herein, your pseudonymized Medical Data may be shared by the Sponsor with different entities both locally and located in other jurisdictions. In addition, your Medical Data may also be transferred to entities located in other jurisdictions for storage and processing purposes.

By signing the present, You expressly consent to the manner in which we will share your pseudonymized Medical Data as well as the international transfer of your pseudonymized Medical Data to the following jurisdictions and entities:

- 6.1.- To Amazon Web Services Company (AWS) with jurisdiction in the United States of America, an international data storage and processing company recognized and used worldwide, where the Sponsor will host the databases in which your pseudonymized Medical Data is stored and processed.
- 6.2. To a laboratory of the Sponsor located in the United Kingdom for the medical-scientific research purposes detailed herein.
- 6.3. To an independent medical professional located in Italy for the medical-scientific research purposes described herein and entrusted by the Sponsor, also for the purpose

of validating the results obtained at the request of the Sponsor, always within the framework of the purposes described herein.

- 6.4. To the Stamboulian Laboratory, a local clinical analysis laboratory owned by CENTRO DE ESTUDIOS INFECTOLÓGICOS SACEI, for the medical-scientific research purposes entrusted by the Sponsor.
- 6.5. To a biobank to be defined by the Sponsor for the purposes foreseen herein and entrusted by the Sponsor. In relation to this point, we inform you that Certain biological samples obtained by virtue of the processes detailed in point 2 herein (also included in the definition of Medical Data), will be stored in a biobank operating within FLENI, or in a biobank belonging to the Sponsor or to a third party designated by the Sponsor, either in Argentina or abroad, for scientific and statistical purposes. In the event that the Sponsor determines that the biobank will be a biobank located abroad, the Sponsor will comply with the legal safeguards required by the applicable regulations regarding the international transfer of its pseudonymized Medical Data.
- 6.6. To other entities to be defined by the Sponsor and always within the framework of the purposes foreseen herein and entrusted by the Sponsor to such entities. In the event that the Sponsor determines to share the data with any other entity, the Sponsor will comply with the legal safeguards required by the applicable regulations in relation to the assignment and/or international transfer of its pseudonymized Medical Data. After the end of the 5-year period covered by the study, the Sponsor of the study may require that the pseudonymized Medical Data be completely anonymized or dissociated from your Identifying Data, and be shared with you, so that such Medical Data will not allow you to be identified. The anonymized Medical Data may then be used by the Sponsor of the study, MULTIPLAI TANGO SAS, for scientific and statistical purposes, without this implying any processing of your Personal Data.

Likewise, once the study is completed, the Center shall keep your Identifying Data and Medical Data for the term established by the applicable regulations, and may only use them for the purposes provided for in such regulations.

In no case will your Identifying Information be published or shared; only the principal investigator of the Center will have access to your Identifying Information and only for the term established by law. Furthermore, your Identifying Information will be kept confidential, even in case of publication of the research results, according to Law Nº 25.326. All study personnel agree to comply with National Law 25.326 on Personal Data Protection. In the future, the information obtained from this study could be used for the development of new research questions.

#### 7. How can I access, modify or delete my personal and genetic data?

In accordance with the provisions of Law No. 25.326, you may at any time access, modify or delete your Identifying Data and/or Medical Data, including blood samples stored in biobanks.

In order to exercise your right to access, update, or rectify, you should contact the Center by sending an e-mail to docencia@lylyk.com.ar. The Center may require you to

identify yourself by asking to see documentation verifying your identity or the information you wish to modify, which will be discarded, if applicable, after verification of the personal data you wish to access.

You may at any time request the Center to delete your Identifying Information and/or Medical Information by sending an e-mail to docencia@lylyk.com.ar. The Center may require you to identify yourself by requesting to see documentation verifying your identity, which will be discarded, if applicable, after verification of the personal data you wish to delete. You should note that certain personal data may not be deleted by the Center under applicable law.

Likewise, you may only exercise your rights of access, updating, rectification and deletion conferred by Law 25.326 against the Center and not against the Sponsor, considering that due to the pseudonymization procedure mentioned in point 6, and the eventual anonymization process also mentioned in point 6, the Sponsor of the study, MULTIPLAI TANGO SAS, will not have at any time, neither during nor after the study, the factual possibility to access, modify or delete your Identifying Data and/or Medical Data.

You accept that the data collected about you that are anonymized will not be susceptible to the exercise of the right of access, modification or deletion, because they are not personal data, since it is not possible to identify you from them.

The Agency for Access to Public Information, the controlling body of Law No. 25,326, is responsible for dealing with complaints and claims filed in relation to non-compliance with the rules on personal data protection.

# 8. Does my participation in the study cost anything and will I receive any compensation for my participation?

No, your participation is voluntary, there is no cost to you and you will not receive any compensation for doing so.

## 9. Who are the researchers in charge of this study?

Dr. Santiago Miriuka as principal investigator and Dr. Gastón Rodríguez Granillo, as principal investigator of the Center. Both will be in charge of the development of the study.

#### 10. Who has evaluated and approved this study?

The present research work has been evaluated and approved by the Clinical Research Ethics Committee (CEIC). If you have any questions about your rights as a participant in a study, please contact us at (5411) 4372-8316, Monday through Friday from 10:00 am to 4:00 pm or by e-mail at info@comitedeeticaceic.com.ar . In the case that an ethical monitoring is carried out at the Center, patients may be summoned with the agreement and authorization of the Principal Investigator (PI), in order to have a conversation about their participation in the study.

#### 11. Who pays for this study?

The budget for the realization of the study will be provided by funds coming exclusively from its Sponsor, MULTIPLAI TANGO SAS. Notwithstanding the foregoing, you are hereby informed that any reference herein to MULTIPLAI TANGO SAS shall also be understood as a reference to MULTIPLAI HEALTH LTD and any other affiliated, controlling or controlled legal entity of the aforementioned legal entities.

## 12. If I have any questions at a later date, or wish to withdraw from the study, how do I do?

| If you have any questions about the study, you may contact the investigators through the following channels of communication: Dr. Santiago Miriuka e-mail: <a href="mailto:santiago@multiplaihealth.com">santiago@multiplaihealth.com</a> Dr. Gastón Rodriguez-Granillo e-mail: <a href="mailto:grodriguezgranillo@gmail.com">grodriguezgranillo@gmail.com</a> | | | |
|---|---|---|---|
| | Having understood the scope o comply with the procedures th participate in the study. | • | |
| | Name of Participant | Date | Participant's signature |
| | Name of Investigator - subinvestigator | Date | Investigator's signature |
| | I have been informed about the | process and purpose of s | toring my biological samples |

□ I voluntarily consent to have my biological samples stored for further unspecified future studies.

□ I "DO NOT" consent to have my blood sample stored.

Date: 06/10/2022 8 Informed Consent -Version 1.1

| Name of Participant | Date | Participant's signature | | | |
|---|---|---|---|---|---|
| | | | Name of Investigator | Date | Investigator's signature |
| | | | G | 2 3.00 | 661.6416. 6 616.1414 |
| - subinvestigator | | | | | |

Informed Consent -Version 1.1 Date: 06/10/2022

9